CLINICAL TRIAL: NCT03259152
Title: Clinical, Pathologic Characteristics and Its Mechansim of Denosumab Treated Giant Cell Tumor of Bone
Brief Title: Characteristics and Mechanism of Denosumab-treated Giant Cell Tumor of Bone
Acronym: D-Gct
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZZ3592-2017
Record Dates: First submitted 2017-08-17; First posted 2017-08-23 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-05

CONDITIONS: Giant Cell Tumor of Bone
Keywords: Giant cell tumor of bone; Denousmab; Pathologic; Clinical; Mechansim
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-Denosumab GctB (Experimental): Specimens obtained during biopsy
  Interventions: Drug: Denosumab
- Post-Denosumab GctB (Experimental): Specimen after administration of Denosumab
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Denosumab (trade names Prolia and Xgeva) is a human monoclonal antibody for the treatment of osteoporosis, treatment-induced bone loss, metastases to bone, and giant cell tumor of bone.Denosumab is a RANKL inhibitor, which works by preventing the development of osteoclasts which are cells that break down bone.
  Other Names: Xgeva or Prolia

SUMMARY:
Giant cell tumor of bone (GCTb) is a primary, osteolytic, benign tumor of the bone. Surgery is the commonly used treatment. Discovery of RANKL and its human monoclonal antibody, denosumab, led to use of denosumab for treatment of GCT. The aim of this study was to evaluate clinical and pathological results of treatment of relapsed or refractoriness GCT with denosumab and to assess adverse effect profile and recurrence rate.

DETAILED DESCRIPTION:
Giant cell tumor of bone (GCTb) is an aggressive, benign bone tumor. GCTb, which was first defined by Cooper and Travers, can produce pulmonary metastasis, albeit rarely (1-6%). GCTb constitutes 5% of primary bone tumors and 20% of benign bone tumors. Histologically, the tumour consists of a proliferation of mononuclear cells, accompanied by a population of non-neoplastic osteoclast-like giant cells and mononuclear osteoclast precursors. Currently, it is thought that proliferating neoplastic cells produce a number of cytokines and mediators, including the receptor activator of nuclear factor κ-B-ligand (RANK-RANKL) system, that recruit osteoclast precursors and induce their maturation into multinucleated osteoclast. The standard management of GCTb is based on surgery with several local adjuvant treatments like methacrylate cement, phenol or cryotherapy to reduce the risk of recurrence, while bisphosphonates are used in some cases to decrease bone resorption and for pain relief in inoperable tumours or metastatic disease. In the last 5 years the use of denosumab, a fully human monoclonal antibody already licensed for postmenopausal osteoporosis and prevention of skeletal related events in bone metastases from solid tumours, has been introduced in the treatment strategy of GCTb. In this study we examined the clinical, radiological, histological and underlying mechanism features of a series of GCTb, before and after denosumab administration, comparing baseline and resection specimens. Moreover, we examined the safety of the drug and on the angiogenesis through the determination of microvascular density (MVD).

ELIGIBILITY:
Inclusion Criteria:

* Giant cell tumor of bone patients confirmed by clinical, medical imaging and Pathology.

Exclusion Criteria:

* (1) less than 14 patients; 2) pregnant patients; 3) A patient who receives other medications during treatment.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Molecular analysis (Immunohistochemistry for RANKL, RANK, OPG,Col-I, VEGF) | 6 month
  For collagen RANKL (Receptor Activator for Nuclear Factor-κ B Ligand), RANK (Receptor Activator for Nuclear Factor-κ B), OPG (Osteoprotegerin), Col-I (type I Collagen), VEGF (Vascular Endothelial Growth Factor) immunohistochemistry, sections were deparaffinized, rehydrated, and immunostained with a SA1024 SABC-POD kit and Kit-0017 DAB detection kit. Briefly, antigen retrieval was performed, and endogenous peroxidases were then inactivated prior to incubation with primary antibodies overnight at 4°C. This was followed by incubation with a biotinylated secondary antibody and a streptavidin-biotin complex peroxidase solution. Diaminobenzidine (DAB) chromogen was applied and counterstained with hematoxylin for antibody detection.
  Images were captured by a microscope system at 400-magnification. The integrated optical density values of each factor were semiquantitatively analyzed using Imaging Pro Plus 6.0 software.
Molecular analysis (RT-PCR for RANKL, RANK, OPG,Col-I, VEGF) | 6 month
  Tissures mRNA was extracted using TRIzol reagent (Invitrogen, Carlsbad, CA). The RNA concentration and quality were assessed using a Quawell Q5000 spectrophotometer (Quawell, San Jose, CA). Reverse transcription PCR was performed using a Gene Amp 7700 Sequence Detection System (Applied Biosystems, Foster City, CA) and custom-designed, validated primers for Col1α1, Col2α1, Aggrecan, MMP-13, and ADAMTS-4. GAPDH was used as the housekeeping gene. Relative gene expression changes were reported using the 2(-Delta Delta C(T)) method as previously described. The experiment was repeated in triplicate to ensure accuracy.

SECONDARY OUTCOMES:
Visual Analog Score - Pain evaluation | 6 months
  Visual analog scale [VAS] is a measure of pain intensity. It is a continuous scale comprised of a horizontal (called horizontal visual analogue scale) or,vertical called vertical visual analog scale usually 10 cm or 100 mm length [both the gradations are used]. It is anchored by two verbal descriptors, one for each symptom extreme. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [on 100-mm scale]
Hematology test - Tartrate Resistant Acid Phosphatase | 6 months
  Tartrate-resistant acid phosphatase, a bone resorption marker, is secreted from osteoclasts and this marker is reported to be high in patients with giant cell tumor of bone. We investigated the effects of denosumab and the usefulness of a tartrate-resistant acid phosphatase as a monitoring marker in the management of a refractory giant cell tumor of bone. Tartrate-resistant acid phosphatase secretion was measured in the patient's serum to monitor the response to denosumab, and a rapid normalization of the marker was observed after the first denosumab administration.
Follow-up for recrudescence | 6 month to 1 year
  Patients were followed up regularly for local or systemic tumor recurrence by X-ray, CT, MRI, ECT.
  The follow-up period was 3 months.
Morphological change - HE (Hematoxylin-Eosin) staining | 6 month
  For histological analysis of the adjacent intervertebral disc and fusion mass, the tissures of the Giant cell tumor of bone were fixed in 10% neutral buffered formalin, decalcified in 10% EDTA-2Na for 3 months, and then embedded in paraffin. They were subsequently cut into 5-mm sections with cationic slides. Slides of the tissures of the Giant cell tumor of bone were stained with H&E and captured by a microscope system (BX53; Olympus, Tokyo, Japan).
Micro-vessel density or area by IHC - stained slides | 6 month
  IHC - stained for VEGF images were used for microvessel density (MVD) and vascular bud relative area analysis. MVD was measured by counting the number of cartilage endplate vascular buds (an average of cephalic and caudal vascular buds). The ratio of vascular bud area to the total endplate area was measured for vascular bud relative area analysis using the grid method. MVD and vascular bud relative area analyses were repeated at least three times for enhanced accuracy
Imaging changes by X-ray, CT, MRI, ECT. | 6 month
  The patients' clinical information, images from radiographs, CT and MRI before and after Denosumab-treatment were recorded and analyzed. Tumor volume was measured on coronal, transverse, and sagital MRI or CT scansof the lesion; and maximum height, width, and depth were recorded; and the volume was calculated using the formula of an ellopsoid mass volume = [(π/6) × height × width × depth]. If CT or MRI were not available, tumor volume was measured on two-plane radiograghs.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 year
  The CTCAE v.4 criteria was used to evaluate late toxicity for all patients. Toxicity scores were recalculated for patients treated before publication of CTCAE v4.0 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuang Zhou, Ph.D, Principal Investigator — Hebei Medical University Third Hospital
Locations (1):
- Zhuang Zhou, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No
We have not yet planned to to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Girolami I, Mancini I, Simoni A, Baldi GG, Simi L, Campanacci D, Beltrami G, Scoccianti G, D'Arienzo A, Capanna R, Franchi A. Denosumab treated giant cell tumour of bone: a morphological, immunohistochemical and molecular analysis of a series. J Clin Pathol. 2016 Mar;69(3):240-7. doi: 10.1136/jclinpath-2015-203248. Epub 2015 Sep 3. PMID 26338802
- [Background] Deveci MA, Paydas S, Gonlusen G, Ozkan C, Bicer OS, Tekin M. Clinical and pathological results of denosumab treatment for giant cell tumors of bone: Prospective study of 14 cases. Acta Orthop Traumatol Turc. 2017 Jan;51(1):1-6. doi: 10.1016/j.aott.2016.03.004. Epub 2016 Oct 24. PMID 27784623
- [Background] Rutkowski P, Ferrari S, Grimer RJ, Stalley PD, Dijkstra SP, Pienkowski A, Vaz G, Wunder JS, Seeger LL, Feng A, Roberts ZJ, Bach BA. Surgical downstaging in an open-label phase II trial of denosumab in patients with giant cell tumor of bone. Ann Surg Oncol. 2015 Sep;22(9):2860-8. doi: 10.1245/s10434-015-4634-9. Epub 2015 Jun 2. PMID 26033180
- See also: Description of Denosumab — https://en.wikipedia.org/wiki/Denosumab